CLINICAL TRIAL: NCT06440655
Title: A Randomized, Split-head Comparison Study of the Efficacy and Safety of Platelet-rich Fibrin and Platelet Rich Plasma in Female Pattern Hair Loss Patients : A Pilot Study
Brief Title: The Efficacy and Safety of Platelet-rich Fibrin and Platelet Rich Plasma in Female Pattern Hair Loss Patients
Acronym: PRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Associate Professor, Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COA no. Si286/2023
Record Dates: First submitted 2024-02-06; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Female Pattern Hair Loss; Platelet-Rich Plasma; Platelet-rich Fibrin
Keywords: female pattern hair loss; platelet-rich plasma; platelet-rich fibrin

STUDY DESIGN:
Intervention Model Description: All subject were injected with PRP and PRF at baseline, 4 weeks and 8 weeks with split-head of sides of injection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRF and PRP (Experimental): All patients were treated with both platelet rich fibrin and platelet rich plasma but each side of head (left or right) was split with
  * one side of head was injected with platelet rich plasma at week 0,4 and 8 (total 3 times)
  * another side of head was injected with platelet rich fibrin at week 0,4 and 8 (total 3 times)
  Interventions: Device: Platelet rich plasma; Device: Platelet rich fibrin

INTERVENTIONS:
Device: Platelet rich plasma — Subjects were treated by Platelet rich plasma in each side of head (Left or right)
  Other Names: PRP
Device: Platelet rich fibrin — Subjects were treated by Platelet rich fibrin in each side of head (Left or right)
  Other Names: PRF

SUMMARY:
The goal of this clinical trial is to compare between platelet-rich fibrin and platelet-rich plasma in female pattern hair loss . The main question[s] it aims to answer are:

* efficacy between platelet-rich fibrin and platelet-rich plasma
* safety between platelet-rich fibrin and platelet-rich plasma Participants will be divided into 2 side of treatment with composed of

  1. Platelet rich plasma
  2. Platelet rich fibrin

DETAILED DESCRIPTION:
Subject was treated both platelet-rich fibrin and platelet-rich plasma for 3 times which 1 month interval then will be followed up at 4 months and 6 months after last treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 20-55 years
* Female
* Subject who was diagnosed with Female pattern hair loss in Ludwig Classification 2 (part width 2-4 centimeters) by Dermatologist

Exclusion Criteria:

* Pregnancy or Lactation subjects
* Subject with history of platelet dysfunction, low platelet, anemia, cirrhosis, cancer, or immunocompromised host
* Subject who are active smoking and alcoholism
* Subject who has dermatitis, scar or infection at intervention area
* Subject who has history of allergy to anesthesia drug
* Subject who taking NSAIDs, Hormonal drug, anticoagulants drug
* Subject who has psychiatric condition diagnosed by psychiatrist
* Subject who are not allowed to take a photo

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Trichoscan | baseline(week0), 4 months after last treatment(week20), 6 months after last treatment(week28)
  Average counts and density of hair per 1.5mm^2

SECONDARY OUTCOMES:
The 7-point of doctor subjective global assessment | baseline(week0),1 month after first treatment(week4), 1 months after second treatment(week8), 4 months after last treatment(week20), 6 months after last treatment(week28)
  Evaluation of improvement through picture by doctor
The 7-point of patient subjective global assessment | baseline(week0),1 month after first treatment(week4), 1 months after second treatment(week8), 4 months after last treatment(week20), 6 months after last treatment(week28)
  Evaluation of improvement through picture by patient
Visual analog scale | baseline(week0), 1 month after first treatment(week4), 1 months after second treatment(week8)
  pain during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rattapon Thuangtong, Asst. Prof., Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok

IPD SHARING:
Plan to Share IPD: No
Prohibited from laws (and/or rules, regulations, contracts). Fear of inappropriate use of data